CLINICAL TRIAL: NCT00986219
Title: A Cross Sectional Study for the Assessment of the Words Used by Patients and Physicians to Express Asthma Symptoms and the Limitations of Daily Activities in Primary Care. The " Asthma Language " Survey
Brief Title: A Study for the Assessment of the Words Used by Patients and Physicians to Express Asthma Symptoms
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-RGR-DUM-2009/1
Record Dates: First submitted 2009-09-22; First posted 2009-09-29 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Asthma
Keywords: Asthma; Language; Symptoms,; Limitation of Daily activities; Patients; Physicians; Greece
MeSH Terms: conditions — Asthma; Language

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asthma Language between patients and physicians

SUMMARY:
The purpose of the study is to evaluate the concordance of the most frequently used words by the patients and the physicians to express asthma symptoms and the limitations of daily activities caused by asthma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of persistent asthma treated with inhaled corticosteroid-based maintenance treatment for at least 6 months and followed up by the investigator for at least the same period of time

Exclusion Criteria:

* Patient with a cardiac disease (congestive heart failure, coronary heart disease)
* Patient with a respiratory disease other than asthma (COPD, sleep apnoea syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care patients with persistent asthma treated with inhaled corticosteroid-based maintenance treatment for at least 6 months and followed up by thep hysician for at least the same period of time.
Sampling Method: Probability Sample
Enrollment: 696 (Actual)
Dates: Start 2009-09; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The concordance of the most frequently used words by the patients and the physicians to express asthma symptoms and the limitations of daily activities caused by asthma | Day 1

SECONDARY OUTCOMES:
The most frequently used words (lexical intensity) by the patient and the physician to express asthma symptoms and the limitations of daily activities. | Day 1
The concordance of words used by physicians and patients according to the level of asthma control (as assessed by ACQ). | Day 1
The actions recommended by the physician or those initiated by the patient and are associated with words that express symptoms. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Mina Gaga, MD, Principal Investigator — Director of the 7th Respiratory Clinic, Sotiria Hospital, Athens, Greece; Panagiotis Pontikis, Dr., Study Director — Marketing Company Medical Director, AstraZeneca Greece
Locations (40):
- Greece (40):
  - Research Site, Pátrai, Achaia
  - Research Site, Agrinio, Aitoloakarnanias
  - Research Site, Thérmo, Aitoloakarnanias
  - Research Site, Naupaktos, Aitoloakarnania
  - Research Site, Argos, Argolida
  - Research Site, Arta, Artas
  - Research Site, Athens, Attica
  - Research Site, Peraious, Attica
  - Research Site, Livadia, Biotias
  - Research Site, Chalcis, Chalkida
  - Research Site, Chalkidiki, Chalkidiki
  - Research Site, Chania, Crete
  - Research Site, Heraklion, Crete
  - Research Site, Rethymno, Crete
  - Research Site, Ermoupoli, Cyclades
  - Research Site, Rhodes, Dodekanisou
  - Research Site, Drama, Drammas
  - Research Site, Kastoria, Florinas
  - Research Site, Amfisa, Fokidos
  - Research Site, Pírgos, Ilia
  - Research Site, Véroia, Imathia
  - Research Site, Ioannina, Ioanninon
  - Research Site, Karditsa, Karditsis
  - Research Site, Chrisoupoli, Kavalas
  - Research Site, Kavala, Kavalas
  - Research Site, Loutraki, Korinthia
  - Research Site, Ptolemaida, Kozani
  - Research Site, Ksanthi, Ksanthis
  - Research Site, Lakonia, Lakonia
  - Research Site, Larissa, Larisas
  - Research Site, Farsala, Larrisa
  - Research Site, Volos, Magnisia
  - Research Site, Kalamata, Messinia
  - Research Site, Katerini, Peierias
  - Research Site, Edessa, Pella
  - Research Site, Komotini, Rodopi
  - Research Site, Serres, Serron
  - Research Site, Igoumenitsa, Thesprotia
  - Research Site, Thessaloniki, Thessalonikis
  - Research Site, Trikala, Trikalon